CLINICAL TRIAL: NCT01812213
Title: Beta-Amyloid Imaging With [18F]NAV4694 Positron Emission Tomography (PET) in Predicting Progression to Alzheimer's Disease (AD) in Subjects With Mild Cognitive Impairment (MCI)
Brief Title: Beta-Amyloid Imaging With [18F]NAV4694 PET in Predicting Progression to AD in Subjects MCI
Acronym: NAV4-04
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Navidea Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NAV4-04
Record Dates: First submitted 2013-03-12; First posted 2013-03-18 (Estimated); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [18F]NAV4694 (Experimental): Intravenous [18F]NAV4694 (8.1 mCi) administered once every 18 months
  Interventions: Drug: [18F]NAV4694

INTERVENTIONS:
Drug: [18F]NAV4694

SUMMARY:
To investigate whether [18F]NAV4694 positron emission tomography (PET) scan findings have the ability to distinguish subjects with mild cognitive impairment (MCI) who progress to Alzheimer's disease (AD) from those who do not.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed informed consent to participate in the study and continues to give willing consent for participation
* Age ≥ 55 years with a diagnosis of MCI
* Educational level of at least 6 years
* Female subjects will not be of child-bearing potential (> 1 year post-menopausal or surgically sterile)
* Availability of a "study partner" who can assist in completing rating scales for the duration of the study
* Cognitive complaints reported by the subject and confirmed by the "study partner"
* Clinical Dementia Rating (CDR) global score = 0.5
* Mini-mental state examination (MMSE) score of 24-30
* Diagnostic and Statistical Manual of Mental Disorders, Version 4, Text Revised (DSM-IV-TR) criteria of dementia not fulfilled

Exclusion Criteria:

* Has been previously enrolled in this study and received the investigational product
* Has received an investigational product within 30 days prior to screening
* Has received disease-modifying therapy that could have changed amyloid brain deposition
* Has exceeded yearly radioactive dose of 30 mSv
* Has a known allergy to the study drug or any of its constituents
* Has a history of alcohol abuse or alcohol dependency in the 3 years prior to study entry, or is an alcoholic or drug addict, as determined by the investigator
* Has ongoing clinically significant (as judged by the investigator), metabolic or any other disease that could currently cause impaired memory (e.g., untreated thyroid disease, vitamin or other nutritional deficiencies, chronic kidney, or liver disease)
* Memory impairment that can be attributed to a disease or condition other than an early phase neurodegenerative syndrome
* Has a parkinsonian movement disorder
* Use of psychoactive medications that would affect the subject's ability to reliably perform neurocognitive testing or create uncertainty in distinguishing between the effects of the psychoactive medication and the subject's underlying cognitive impairment (e.g., benzodiazepines, sedatives, antipsychotics)
* Has received any contrast material (X-ray, MRI) or radiopharmaceutical within 48 hours prior to, or a therapeutic radiopharmaceutical (e.g., 131I) within 10 days prior to, or any radiopharmaceutical administration within 10 radioactive half-lives prior to the administration of the investigational product or for whom administration of such substances is planned within 7 days after investigational product administration
* History of major recurrent depressive disorder (per DSM-IV-TR) within the last 5 years prior to screening
* Has a brain tumor or other intracranial lesion, a disturbance of cerebral spinal fluid circulation (e.g., normal pressure hydrocephalus), and/or a significant history of head trauma or brain surgery
* Has signs of major cerebrovascular disease, as verified by medical history and/or brain MRI
* Is scheduled for surgery and/or another invasive procedure within the 7 days following investigational product administration
* Has any contraindication to MRI examination, e.g., metal implants, phobia, or cannot undergo an MRI for other reasons such as the inability to lie flat

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Reininger, MD, PhD, Study Director — Navidea Biopharmaceuticals Inc.
Locations (11):
- United States (11):
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Galiz Research, Hialeah, Florida
  - Mt. Sinai Wien Center for Alzheimer's Disease, Miami Beach, Florida
  - Compass Research, Orlando, Florida
  - Rush University Medical Center, Chicago, Illinois
  - SIU School of Medicine, Springfield, Illinois
  - McLean Hospital, Belmont, Massachusetts
  - Qunicy Medical Center, Alzheimer's Disease Center, Quincy, Massachusetts
  - Neurological Associates of Albany, Albany, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Wake Forest School of Medicine, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- [18F]NAV4694: Intravenous [18F]NAV4694 (8.1 mCi) administered once every 18 months
  [18F]NAV4694
Period: Overall Study
Arm/Group | [18F]NAV4694
Started | 76
Completed | 39
Not Completed | 37

BASELINE CHARACTERISTICS:
Arm/Group | [18F]NAV4694
Number analyzed (Participants) | 76
Age, Continuous [Mean (Full Range); unit: years] | 76 [59 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 66
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 72
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Mild Cognitive Impairment Progression to Alzheimer's Disease
Description: Incidence of Mild Cognitive Impairment Progression to Alzheimer's Disease
Time Frame: 3 Years
Population: Trial terminated prior to collection of sufficient information to evaluate the outcome measure. Data not collected.
Arm/Group | [18F]NAV4694
Number analyzed (Participants) | 0

2. Secondary Outcome: Incidence of [18F]NAV4694 PET Positive Scans at 18 Months Compared to Baseline
Description: Incidence of [18F]NAV4694 PET Positive scans at 18 months compared to baseline
Time Frame: 18 months
Population: Trial terminated prior to collection of sufficient information to evaluate the outcome measure. Data not collected.
Arm/Group | [18F]NAV4694
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Neuro-cognitive Test Battery Scores at 6 Months Compared to Baseline
Description: Change in Neuro-cognitive Test Battery Scores at 6 months compared to baseline
Time Frame: 6 months
Population: Trial terminated prior to collection of sufficient information to evaluate the outcome measure. Data not collected.
Arm/Group | [18F]NAV4694
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Neuro-cognitive Test Battery Scores at 12 Months Compared to Baseline
Description: Change in Neuro-cognitive Test Battery Scores at 12 months compared to baseline
Time Frame: 12 months
Population: Trial terminated prior to collection of sufficient information to evaluate the outcome measure. Data not collected.
Arm/Group | [18F]NAV4694
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Neuro-cognitive Test Battery Scores at 18 Months Compared to Baseline
Description: Change in Neuro-cognitive Test Battery Scores at 18 months compared to baseline
Time Frame: 18 months
Population: Trial terminated prior to collection of sufficient information to evaluate the outcome measure. Data not collected.
Arm/Group | [18F]NAV4694
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in Neuro-cognitive Test Battery Scores at 24 Months Compared to Baseline
Description: Change in Neuro-cognitive Test Battery Scores at 24 months compared to baseline
Time Frame: 24 months
Population: Trial terminated prior to collection of sufficient information to evaluate the outcome measure. Data not collected.
Arm/Group | [18F]NAV4694
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in Neuro-cognitive Test Battery Scores at 30 Months Compared to Baseline
Description: Change in Neuro-cognitive Test Battery Scores at 30 months compared to baseline
Time Frame: 30 months
Population: Trial terminated prior to collection of sufficient information to evaluate the outcome measure. Data not collected.
Arm/Group | [18F]NAV4694
Number analyzed (Participants) | 0

8. Secondary Outcome: Change in Neuro-cognitive Test Battery Scores at 36 Months Compared to Baseline
Description: Change in Neuro-cognitive Test Battery Scores at 36 months compared to baseline
Time Frame: 36 months
Population: Trial terminated prior to collection of sufficient information to evaluate the outcome measure. Data not collected.
Arm/Group | [18F]NAV4694
Number analyzed (Participants) | 0

9. Secondary Outcome: Change in SUVR Scores at 18 Months Compared to Baseline
Description: Change in SUVR scores at 18 months compared to baseline
Time Frame: 36 months
Population: Trial terminated prior to collection of sufficient information to evaluate the outcome measure. Data not collected.
Arm/Group | [18F]NAV4694
Number analyzed (Participants) | 0

10. Secondary Outcome: Incidence of Adverse Events Post Baseline
Description: Incidence of Adverse Events post baseline
Time Frame: 3 Years
Population: All participants
Measure: Number; unit: Post-baseline adverse events
Arm/Group | [18F]NAV4694
Number analyzed (Participants) | 76
Post-baseline adverse events | 43

ADVERSE EVENTS:
Time Frame: Up to 36 months
Arm/Group | [18F]NAV4694
All-Cause Mortality (participants affected / at risk) | 0/76
Serious Adverse Events (participants affected / at risk) | 14/76
Other Adverse Events (participants affected / at risk) | 16/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [18F]NAV4694 (N=76)
Cardiac failure congestive (Cardiac disorders) | 1 (2)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2)
Post Laminectomy Syndrome (Injury, poisoning and procedural complications) | 1 (1)
Meningitis bacterial (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Cervical vertebral fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung carcinoma cell type unspecified stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Colon cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [18F]NAV4694 (N=76)
Nausea (Gastrointestinal disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Systolic hypertension (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Medication error (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Fatigue (General disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT01812213/Prot_SAP_000.pdf